CLINICAL TRIAL: NCT01023555
Title: Increasing the Yield of Blood Cultures in the Neonatal Intensive Care Unit- A Prospective Controlled Trial
Brief Title: Increasing the Yield of Blood Cultures in Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Ruben Bromiker MD, Shaare Zedec Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: SZMC-bromi
Record Dates: First submitted 2009-12-01; First posted 2009-12-02 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Bacteremia
Keywords: Bacteremia; Blood Cultures; Sepsis
MeSH Terms: conditions — Bacteremia; Sepsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5cc 2 Bottles (No Intervention)
- 1cc single bottle (Active Comparator)
  Interventions: Other: 1cc of blood in a single aerobic culture bottle

INTERVENTIONS:
Other: 1cc of blood in a single aerobic culture bottle — The efficacy of using 1cc of blood in a single aerobic bottle for cultures in neonatal bacteremia will will be compared with the traditional 0.5cc of blood in 2 Bottles
  Arms: 1cc single bottle

SUMMARY:
The purpose of this study is to determine whether the use of a single blood sample of 1cc in an aerobic bottle will provide a better yield and time to positivity than 2 samples of 0.5 cc in 2 (aerobic and anaerobic) bottles for blood cultures in neonates.

ELIGIBILITY:
Inclusion Criteria:

* All blood cultures taken in the NICU during the study period.

Exclusion Criteria:

* Bacteria that are normal flora of the skin such as Coagulase negative staphylococci or Streptococci Viridans are considered, except if grown in two sets of cultures or in the presence of laboratory and clinical indices of infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Non Inferiority of 1 cc blood culture in a single aerobic bottle instead of 0.5 cc for 2 bottles. | 6months

SECONDARY OUTCOMES:
utility of the routine use of anaerobic bottle for blood cultures in newborns | 6 months
Comparison of time to positivity of 1 cc blood culture in a single aerobic bottle instead of 0.5 cc for 2 bottles (aerobic and anaerobic) | 6 months

REFERENCES:
- [Derived] Yaacobi N, Bar-Meir M, Shchors I, Bromiker R. A prospective controlled trial of the optimal volume for neonatal blood cultures. Pediatr Infect Dis J. 2015 Apr;34(4):351-4. doi: 10.1097/INF.0000000000000594. PMID 25764096